CLINICAL TRIAL: NCT01567020
Title: Central Auditory Processing Deficits Associated With Blast Exposure
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C7755-I
Record Dates: First submitted 2012-03-02; First posted 2012-03-30 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Blast Injuries; Brain Injuries; Age Factors
Keywords: Central Auditory Processing; Traumatic Brain Injury; Hearing Loss
MeSH Terms: conditions — Blast Injuries; Brain Injuries; Brain Injuries, Traumatic; Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Biospecimen Retention: None Retained — None collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control: Non-blast-exposed and non-TBI, aged younger than 50
  Interventions: Other: Diagnostic
- Blast: Blast-exposed with or without a TBI diagnosis
  Interventions: Other: Diagnostic
- Non-Blast-Exposed TBI: Non-blast-exposed with TBI diagnosis
  Interventions: Other: Diagnostic
- Older: Non-blast-exposed and non-TBI, aged 50 or older
  Interventions: Other: Diagnostic

INTERVENTIONS:
Other: Diagnostic — All participants will be evaluated with a battery of behavioral and electrophysiological measures to assess central auditory processing abilities.

SUMMARY:
The current conflicts in Afghanistan and Iraq have resulted in unprecedented rates of exposure to high-intensity blasts and resulting brain injury. This research team has established that recently blast-exposed Soldiers show differences from controls on tests of central auditory function. This project will 1) develop a more accurate estimate of the prevalence of central auditory dysfunction among Veterans exposed to blasts over the past ten years, 2) identify the functional outcomes associated with abnormal performance on tests of central processing, and 3) improve understanding of the ways in which blast-exposure resembles and differs from both the normal aging process and non-blast-related TBI in terms of performance on tests of central auditory processing.

DETAILED DESCRIPTION:
The current conflicts in Afghanistan (Operation Enduring Freedom; OEF) and Iraq (Operation Iraqi Freedom; OIF) have resulted in unprecedented rates of exposure to high-intensity blasts and resulting brain injury. Dennis (2009) reports that during 2005-2007, 68% of U.S. military personnel injured in the OEF/OIF conflicts had blast-related injuries and 28%-31% of those evacuated to Walter Reed Army Medical Center (WRAMC), Washington, DC had brain injuries. While the common focus of auditory evaluation is on damage to the peripheral auditory system, the prevalence of brain injury among those exposed to high-intensity blasts suggests that damage to the central auditory system is an equally important concern for the blast-exposed Veteran. Discussions with clinical audiologists and OEF/OIF Veterans Service Office personnel suggest that a common complaint voiced by blast-exposed Veterans is an inability to understand speech in noisy environments, even when peripheral hearing is within normal or near-normal limits (see attached letters of support). Such complaints are consistent with damage to neural networks responsible for higher-order auditory processing. This proposal is the second phase of a research project focused on examining the degree to which central auditory processing (CAP) dysfunction is a result of blast exposure. Over the initial period of funding, data collection at WRAMC and the VA RR&D National Center for Rehabilitative Auditory Research (NCRAR) established that CAP dysfunction is present in Warfighters exposed to high-intensity blasts while serving in combat. Recently blast-exposed patients with and without diagnoses of mild traumatic brain injury (mTBI) tested at WRAMC showed differences from controls tested at NCRAR on one or more behavioral and neurophysiological tests used to evaluate central auditory function. This project will 1) develop a more accurate estimate of the prevalence of central auditory dysfunction among Veterans exposed to blasts over the past ten years, 2) identify the functional outcomes associated with abnormal performance on tests of central processing, and 3) improve understanding of the ways in which blast-exposure resembles and differs from both the normal aging process and non-blast-related TBI in terms of performance on tests of central auditory processing.

Key Question 1: To what extent is CAP dysfunction observable among OEF/OIF Veterans who have been exposed to high intensity blasts? Based on preliminary data, the investigators hypothesize that the rate of abnormal performance on behavioral and neurophysiological tests of CAP dysfunction will be higher in a group of Veterans exposed to blasts than it will be in a control group of similar ages and hearing thresholds who have not been exposed to blasts.

Key Question 2: How well can behavioral and neurophysiological tests of CAP predict functional auditory deficits measured behaviorally and through self report? It is hypothesized that tests of CAP ability will predict performance in a testing situation involving multiple talkers delivering competing messages. CAP tests will also correlate with responses blast-exposed Veterans make on the Speech and Spatial Qualities of Hearing (SSQ) questionnaire, designed to examine functional hearing ability in various acoustically complex environments.

Key Question 3: To what extent do blast-exposed Veterans resemble older listeners and participants with mild TBI who have not been exposed to blasts in their performance on CAP tests and functional tests of hearing? It is hypothesized that comparisons of the blast-exposed group with an older group with matched pure-tone sensitivity and an age- and hearing-matched group with non-blast-related TBI will be consistent with premature aging in the blast-exposed group but demonstrate substantive differences with the non-blast group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90
* Pure-tone sensitivity of 40 dB HL or better at all audiometric frequencies below 8 kHz
* English as first language.

Group membership inclusion criteria:

Group 1: Blast exposed Veterans

* Report having been exposed to high-intensity blast during the ten years prior to enrollment
* Cognitive and physical ability to take part in these auditory evaluations

Group 2. Non-blast TBI group

* Diagnosed with mild-to-moderate TBI

Group 3. Age matched control group -18-59 years.

Group 4. Older control group

* 60-90 years.
* Older group will be aged 60 and older

Audiometric status of these groups will be required to meet the same exclusion criteria as that of the other two groups described above

Exclusion Criteria:

* Evidence of conductive or retrocochlear dysfunction
* Hearing loss exceeding pure-tone averages for frequencies of .5, 1, 2, and 4 kHz of 35 dB HL

  --Hearing loss of greater than 40 dB HL at any one of these frequencies in either ear
* Asymmetrical hearing thresholds exceeding 10 dB at any audiometric frequency below 4 kHz
* Abnormal cognitive function as indicated by scores of 23 or below on the Mini Mental State Exam
* Indications of clinical depression as evidenced by a score of 17 or greater on the Beck Depression Inventory

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick J Gallun, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be through an established data repository overseen by the VA Portland HCS IRB.
Supporting Information: Analytic Code
Time Frame: Available starting Jan 2016, and continuing to be available as long as a repository director is available to oversee the data.
Access Criteria: IRB approved protocol allowing data to be transferred from repository to recipient study.

REFERENCES:
- [Background] Fausti SA, Wilmington DJ, Gallun FJ, Myers PJ, Henry JA. Auditory and vestibular dysfunction associated with blast-related traumatic brain injury. J Rehabil Res Dev. 2009;46(6):797-810. doi: 10.1682/jrrd.2008.09.0118. PMID 20104403

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older
Started | 28 | 46 | 20 | 11
Completed | 21 | 41 | 18 | 10
Not Completed | 7 | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older | Total
Number analyzed (Participants) | 21 | 41 | 18 | 10 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 41 | 18 | 8 | 88
  >=65 years | 0 | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.5) | 38.4 (11.8) | 40.4 (10.9) | 56.4 (5.5) | 38.82 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 2 | 3 | 14
  Male | 14 | 39 | 16 | 7 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 41 | 18 | 10 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Blast-exposed Veterans With Abnormal Abilities in One or More Behavioral Tests of Central Auditory Processing
Description: Tests to be administered:
  Dichotic Digits Test: Percentage of digits reported correctly from 0 (worst performance) to 100 (best performance) Gaps in Noise Test: Approximate threshold in milliseconds from 2 (best) to 20 (worst) Staggered Spondaic Words Test: Total number of errors from 0 (best) to 40 (worst) Masking Level Differences Test: Difference in threshold between diotic and dichotic stimuli in decibels from 0 (worst) to 24 (best) Frequency Pattern Test: Percentage of sequences reported correctly from 0 (worst performance) to 100 (best performance) Adaptive Tests of Temporal Resolution: Not reported due to software error in stimulus presentation
Time Frame: six months
Population: Note that some of the participants finished all of the primary outcome measures but withdrew without finishing all of the secondary tests. They are thus listed as having withdrawn but are still included here for completeness.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older
Number analyzed (Participants) | 22 | 42 | 14 | 11
units on a scale
  Dichotic Digits (RE) | 99.1 (1.23) | 95.2 (5.5) | 96.6 (3.3) | 97.5 (3.2)
  Gaps in Noise (RE) | 4.7 (1.1) | 6.4 (2.2) | 5.6 (1.7) | 4.7 (1.5)
  Staggerred Spondaic Words (Total Errors) | 2.1 (1.8) | 7.9 (7.7) | 5 (6.04) | 4.1 (2.4)
  Frequency Pattern Test (RE) | 95.5 (8.6) | 86.8 (15.5) | 84.3 (21.1) | 90.3 (10.8)
  Masking Level Difference | 13.4 (2.9) | 12.1 (2.5) | 12 (2.4) | 9.8 (2.8)

2. Secondary Outcome: Ratings of Self-reported Ability to Process Auditory Information in Various Settings
Description: Hearing Health Inventory for Adults is a 25 item questionnaire that asks participants to rank how often auditory issues create problems in daily life. Scores range from 0 to 100, with higher scores indicating greater perceived levels of handicap.
Time Frame: six months
Population: Not all participants were available for further testing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older
Number analyzed (Participants) | 13 | 16 | 0 | 0
score on a scale | 6.75 (12.8) | 32.5 (31.33) |  |

3. Secondary Outcome: Functional Hearing Ability in Multitalker Environments
Description: The Functional Hearing Questionnaire (FHQ), developed for veterans with brain injuries was used to evaluate self perceived hearing difficulties. The FHQ is a nine item questionnaire that asks participants to rate their level of difficulty hearing in different circumstances on a four point scale. Scores range from 9 to 36, with higher scores indicating a greater level of difficulty.
Time Frame: six months
Population: Not all participants were available for further testing.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older
Number analyzed (Participants) | 13 | 16 | 0 | 0
scores on a scale | 15.2 (3.9) | 19.9 (6.1) |  |

4. Secondary Outcome: Percent Change in P2 Component of Electrophysiological Response
Description: Average change in amplitude of the P2 component of the electrophysiological response to paired clicks. Habituation to the clicks is anticipated, resulting in a large percentage change in amplitude to the second click.
Time Frame: six months
Population: This analysis was only conducted on a subset of the sample, as not all were available for further testing.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older
Number analyzed (Participants) | 16 | 13 | 0 | 0
Percent Change | 65.74 (13.8) | 51.87 (16) |  |

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Control | Blast | Non-Blast-Exposed TBI | Older
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/46 | 0/20 | 0/11
Other Adverse Events (participants affected / at risk) | 0/28 | 0/46 | 0/20 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes